CLINICAL TRIAL: NCT02500056
Title: Single-centre Single-blinded Randomised Study Evaluating the Impact of Mesh Pore Size on Chronic Pain After Lichtenstein Hernioplasty
Brief Title: Study Evaluating the Impact of Mesh Pore Size on Chronic Pain After Lichtenstein Hernioplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tartu University Hospital (Other)
Responsible Party: Principal Investigator, Ceith Nikkolo, Dr., Tartu University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10100
Record Dates: First submitted 2015-07-10; First posted 2015-07-16 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Inguinal Hernia
Keywords: Inguinal hernia; Chronic pain; Mesh; Lichtenstein hernioplasty
MeSH Terms: conditions — Hernia, Inguinal; Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- OM group (Active Comparator): Optilene LP mesh
  Interventions: Device: Optilene LP mesh
- UM group (Active Comparator): Ultrapro mesh
  Interventions: Device: Ultrapro mesh

INTERVENTIONS:
Device: Optilene LP mesh — Lichtenstein hernioplasty
  Arms: OM group
Device: Ultrapro mesh — Lichtenstein hernioplasty
  Arms: UM group

SUMMARY:
The aim of the present study is to determine whether usage of mesh with larger pores, compared with mesh with smaller pores, would result in decreased rate of chronic pain after open inguinal hernia repair.

DETAILED DESCRIPTION:
The aim of the present study is to determine whether usage of mesh with larger pores, compared with mesh with smaller pores, would result in decreased rate of chronic pain after open inguinal hernia repair. The patients are randomized into two study gropus receiving mesh with different pore size. Clinical follow-up examination will be performed 1 week, 1 month, 6 months and 3 years after the operation.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* unilateral primary reducible inguinal hernia
* elective operation
* consent to participate in the study.

Exclusion Criteria:

* age <18 years
* irreducible
* strangulated
* recurrent hernia
* inability to understand the questionnaire
* unwillingness to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2015-04 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OM Group | UM Group
Started | 70 | 73
Completed | 63 | 65
Not Completed | 7 | 8
Not completed — Lost to Follow-up | 3 | 7
Not completed — Recurrence | 1 | 0
Not completed — Death | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OM Group | UM Group | Total
Number analyzed (Participants) | 63 | 65 | 128
Age, Customized [Number; unit: participants] — >=18 years
  participants
    >=18 years | 63 | 65 | 128
Sex/Gender, Customized [Number; unit: participants] — Gender (male + female)
  participants
    Female | 3 | 10 | 13
    Male | 60 | 55 | 115
Unilateral inguinal hernia [Number; unit: participants] | 63 | 65 | 128
Primary inguinal hernia [Number; unit: participants] | 63 | 65 | 128
Reducible inguinal hernia [Number; unit: participants] | 63 | 65 | 128
Elective operation [Number; unit: participants] | 63 | 65 | 128

OUTCOME MEASURES:

1. Primary Outcome: Chronic Pain
Description: On visual analogue scale pain measurement at rest, on coughing, when rising from lying to sitting and during physical effort and exercise
Time Frame: 6-month follow-up
Measure: Number; unit: percentage of patients with pain
Arm/Group | OM Group | UM Group
Number analyzed (Participants) | 67 | 67
percentage of patients with pain | 34.3 | 46.3

2. Secondary Outcome: Chronic Pain
Description: as for outcome 1
Time Frame: 3-year follow-up
Measure: Number; unit: percentage of patients with pain
Arm/Group | OM Group | UM Group
Number analyzed (Participants) | 63 | 65
percentage of patients with pain | 15.9 | 33.9

3. Secondary Outcome: Foreign Body Feeling
Description: The question about foreign body feeling was a yes-or-no question
Time Frame: 6-month follow-up
Population: Drop-outs at 6-month follow-up (3+6) not included
Measure: Number; unit: percentage of patients with foreign body
Arm/Group | OM Group | UM Group
Number analyzed (Participants) | 67 | 67
percentage of patients with foreign body | 31.3 | 47.8

ADVERSE EVENTS:
Time Frame: 3-year
Arm/Group | OM Group | UM Group
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/65
Other Adverse Events (participants affected / at risk) | 10/63 | 10/65
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OM Group (N=63) | UM Group (N=65)
Seroma (Surgical and medical procedures) | 2 (2) | 1 (1)
Haematoma (Surgical and medical procedures) | 8 (8) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No